CLINICAL TRIAL: NCT04503421
Title: Use of Blood Flow Restriction (BFR) Therapy in Post-operative Rehabilitation Following Distal: A Prospective Randomized Control Trial
Brief Title: Use of Blood Flow Restriction (BFR) Therapy in Post-operative Rehabilitation Following Distal Biceps Tendon Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Charles S Day, Orthopedic Surgeon, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Henry - IRB00000253
Record Dates: First submitted 2020-07-28; First posted 2020-08-07 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Bicep Tendon Rupture
Keywords: blood flow restriction; Rehabilitation; Physical therapy
MeSH Terms: interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BFR (Experimental): Patient will use the following rehabilitation protocol while incorporating blood flow restriction therapy:
  * Post-op weeks 0-6: Passive shoulder and wrist Range of Motion (ROM) only
    * Sling immobilization with active wrist and shoulder ROM
    * Active extension of biceps to 30 degrees, No active flexion
  * 6-9 weeks full active extension in brace
    * Maintain wrist and shoulder flexibility
    * Begin rotator cuff/deltoid isometrics, progress active extension in brace
  * Weeks 9-12: Gently advance ROM to tolerance
    * Discontinue sling
    * Begin active flexion and extension against gravity.
    * Advance strength to light resistance, maintain flexibility/ROM
  * Weeks 12-6 months: Gradual return to full ROM and pain free o Begin gradual flexion strengthening and advance as tolerated
  Interventions: Other: Blood Flow Restriction Therapy
- Control (no BFR) (No Intervention): patients will use following rehabilitation protocol without the use of blood flow restriction therapy:
  * Post-op weeks 0-6: Passive shoulder and wrist Range of Motion (ROM) only
    * Sling immobilization with active wrist and shoulder ROM
    * Active extension of biceps to 30 degrees, No active flexion
  * 6-9 weeks full active extension in brace
    * Maintain wrist and shoulder flexibility
    * Begin rotator cuff/deltoid isometrics, progress active extension in brace
  * Weeks 9-12: Gently advance ROM to tolerance
    * Discontinue sling
    * Begin active flexion and extension against gravity.
    * Advance strength to light resistance, maintain flexibility/ROM
  * Weeks 12-6 months: Gradual return to full ROM and pain free o Begin gradual flexion strengthening and advance as tolerated

INTERVENTIONS:
Other: Blood Flow Restriction Therapy — Use of a tourniquet set to 50% of limb occlusion pressure while performing post operative physical therapy
  Arms: BFR

SUMMARY:
The goal of this investigation is to determine if using BFR during postoperative therapy would lead to increased and expedited strength gains. Additionally, the investigators would like to determine if BFR is beneficial in preventing muscle atrophy and fatty infiltration in the setting of bicep tendon tears, due to the altered tension-length relationship following surgery. The study will also look at patient reported outcomes metrics and pain scores to determine if BFR has a significant impact on the patient experience surrounding distal biceps tear and surgical repair

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* Undergoing distal biceps tendon repair

Exclusion Criteria:

* Revision Biceps tendon repair,
* Irrepairable tendon injury,
* Biceps repairs with biologic augmentation,
* Patients with concomitant neurovascular injury,
* Inability to tolerate BFR treatment,
* Unable to complete full course of physical therapy,
* Peripheral vascular disease,
* History of Venous thromboembolism (VTE)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Strength | 1 week post-operatively
  measured via dynamometer (pounds)
Strength | 6 weeks post-operatively
  measured via dynamometer (pounds)
Strength | 3 months post-operatively
  measured via dynamometer (pounds)
Strength | 6 months post-operatively
  measured via dynamometer (pounds)

SECONDARY OUTCOMES:
Range of Motion | 1 week post-operatively
  via goniometer (degrees)
Range of Motion | 6 week post-operatively
  via goniometer (degrees)
Range of Motion | 3 months post-operatively
  via goniometer (degrees)
Range of Motion | 6 months post-operatively
  via goniometer (degrees)
Perceived Pain | 1 week post-operatively
  via visual analog scale (VAS) pain scale: (scale 0 - 10, higher score indicates more pain)
Perceived Pain | 6 week post-operatively
  via visual analog scale (VAS) pain scale: (scale 0 - 10, higher score indicates more pain)
Perceived Pain | 3 months post-operatively
  via visual analog scale (VAS) pain scale: (scale 0 - 10, higher score indicates more pain)
Perceived Pain | 6 months post-operatively
  via visual analog scale (VAS) pain scale: (scale 0 - 10, higher score indicates more pain)
Patient reported outcome scores | 1 week post-operatively
  via Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function (PF) score
Patient reported outcome scores | 1 week post-operatively
  via Patient-Reported Outcomes Measurement Information System (PROMIS) Pain (P) score
Patient reported outcome scores | 1 week post-operatively
  via Patient-Reported Outcomes Measurement Information System (PROMIS) Depression (D) score
Patient reported outcome scores | 6 week post-operatively
  via Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function (PF) score
Patient reported outcome scores | 6 week post-operatively
  via Patient-Reported Outcomes Measurement Information System (PROMIS) Pain (P) score
Patient reported outcome scores | 6 week post-operatively
  via Patient-Reported Outcomes Measurement Information System (PROMIS) Depression (D) score
Patient reported outcome scores | 3 months post-operatively
  via Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function (PF) score
Patient reported outcome scores | 3 months post-operatively
  via Patient-Reported Outcomes Measurement Information System (PROMIS) Pain (P) score
Patient reported outcome scores | 3 months post-operatively
  via Patient-Reported Outcomes Measurement Information System (PROMIS) Depression (D) score
Patient reported outcome scores | 6 months post-operatively
  via Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function (PF) score
Patient reported outcome scores | 6 months post-operatively
  via Patient-Reported Outcomes Measurement Information System (PROMIS) Pain (P) score
Patient reported outcome scores | 6 months post-operatively
  via Patient-Reported Outcomes Measurement Information System (PROMIS) Depression (D) score

CONTACTS AND LOCATIONS:
Locations (1):
- Health Ford Health System, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wernbom M, Augustsson J, Raastad T. Ischemic strength training: a low-load alternative to heavy resistance exercise? Scand J Med Sci Sports. 2008 Aug;18(4):401-16. doi: 10.1111/j.1600-0838.2008.00788.x. Epub 2008 May 3. PMID 18466185
- [Background] Huynh T, Leiter J, MacDonald PB, Dubberley J, Stranges G, Old J, Marsh J. Outcomes and Complications After Repair of Complete Distal Biceps Tendon Rupture with the Cortical Button Technique. JB JS Open Access. 2019 Aug 27;4(3):e0013.1-6. doi: 10.2106/JBJS.OA.19.00013. eCollection 2019 Jul-Sep. PMID 31592499
- [Background] Ohta H, Kurosawa H, Ikeda H, Iwase Y, Satou N, Nakamura S. Low-load resistance muscular training with moderate restriction of blood flow after anterior cruciate ligament reconstruction. Acta Orthop Scand. 2003 Feb;74(1):62-8. doi: 10.1080/00016470310013680. PMID 12635796
- [Background] Takarada Y, Takazawa H, Ishii N. Applications of vascular occlusion diminish disuse atrophy of knee extensor muscles. Med Sci Sports Exerc. 2000 Dec;32(12):2035-9. doi: 10.1097/00005768-200012000-00011. PMID 11128848
- [Background] Clark BC, Manini TM, Hoffman RL, Williams PS, Guiler MK, Knutson MJ, McGlynn ML, Kushnick MR. Relative safety of 4 weeks of blood flow-restricted resistance exercise in young, healthy adults. Scand J Med Sci Sports. 2011 Oct;21(5):653-62. doi: 10.1111/j.1600-0838.2010.01100.x. Epub 2010 Mar 11. PMID 21917016